CLINICAL TRIAL: NCT05423938
Title: Efficacy of Two Formulas of Oral Nutritional Supplementation on Metabolic Parameters and Glycemic Monitoring in Patients at Nutritional Risk With Type 2 Diabetes Mellitus
Brief Title: Efficacy of Two ONS in Patients at Nutritional Risk With Type 2 Diabetes Mellitus
Acronym: DIACARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Collaborators: Adventia Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DIACARE
Record Dates: First submitted 2022-06-14; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Type 2 Diabetes; Malnutrition
Keywords: ONS; Type 2 diabetes; Malnutrition; EVOO; carbohydrates; glycemic index
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Malnutrition | interventions — Diet, Diabetic

STUDY DESIGN:
Intervention Model Description: Randomized, crossover, double blind, multicenter, clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bi1 diacare hp-hc (Experimental): During 6 days, patients received 2 ONS of a specific formula for diabetes, high energy (300 kcal/unit) and high protein (20%), with fiber, EPA&DHA, EVOO and a specific mix of low glycemic index of carbohydrate
  Interventions: Dietary Supplement: Diabetic
- Control (Active Comparator): During 6 days, patients received 2 ONS of a standar formula, high energy (300 kcal/unit) and high protein (20%), without fiber, without EPA&DHA, without EVOO and without a specific mix of low glycemic index of carbohydrate
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Diabetic — It is a hypercaloric and hyperproteic dietary supplement formulated to contribute to control the glycemia with: a specific mix of carbohydrate with a low GI, fiber, EVOO and EPA&DHA
  Other Names: Bi1 diacare hp-hc
  Arms: Bi1 diacare hp-hc
Dietary Supplement: Control — It is a hypercaloric and hyperproteic dietary supplement formulated without the ingredients to contribute in the glycemia control
  Arms: Control

SUMMARY:
Rationale: The aim of the study was to compare the glycemic and insulinemic response of malnourished patients with type 2 diabetes after oral feed between a diabetic oral nutritional supplements (ONS) and a standard one.

Methods: Randomized, double-blind, crossover, multicenter clinical trial, conducted in patients with type 2 diabetes and a diagnosis of malnutrition (SGA). Patients were randomized to receive two ONS: diabetic (Bi1 diacare hp/hc) or control (standard, isocaloric and isoproteic), a week apart. A glycemia and insulinemia curve was made at times: 0', 30', 60', 90', 120', and 180', after drank 200 ml of the ONS. The analyzed variables were the area under the curve (AUC 0-t) of glucosa and insulin, and the maximum concentration of glucose (Cmax).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with DM2 (confirmed by the use of oral hypoglycemic agents for at least two months).
* Patients at nutritional risk diagnosed through the Subjective Global Assessment.
* Adequate cultural level and understanding of the clinical study.
* Agree to voluntarily participate in the study and give their informed consent in writing.
* Non-pregnant and non-lactating women or women who have given birth at least six weeks prior to the screening visit.

Exclusion Criteria:

1. Type 1 DM, DM2 with insulin treatment and DM secondary to steroids.
2. Consumption of alpha-glucosidase inhibitors.
3. Current infection (requiring medication or hospitalization), patients undergoing inpatient surgery, or receiving corticosteroids within the past three months or antibiotics within the past three weeks prior to Screening Visit.
4. BMI > 35 Kg/m2.
5. Active malignant neoplasm (except the following dermal malignancies: basal cell carcinoma, squamous cell carcinoma, carcinoma in situ of the cervix uteri).
6. End-stage organ failure (such as end-stage renal disease) or organ transplant.
7. Advanced chronic kidney disease (glomerular filtration rate < 30 ml/min).
8. Severe liver disease.
9. Severe gastroparesis.
10. Chronic infectious disease, such as active tuberculosis, hepatitis B or C, or HIV infection.
11. Consumption of phytotherapy products, dietary supplements or medications except oral hypoglycemic agents, during the four weeks prior to the screening visit, which could profoundly affect (in the opinion of the PI) blood glucose.
12. Allergy or intolerance to any component of the products under study.
13. Participation in a concurrent trial that conflicts with this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2022-02-17 (Actual)

PRIMARY OUTCOMES:
Postprandial glycemic response | 180 minutes

SECONDARY OUTCOMES:
Postprandial insulin response | 180 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- José M. García Almeida, Málaga, Spain

IPD SHARING:
Plan to Share IPD: No